CLINICAL TRIAL: NCT02210377
Title: Department of Traditional Chinese Medicine, Kaohsiung Chang Gung Memorial Hospital and Chang Gung University College of Medicine, Kaohsiung
Brief Title: A Preliminary Randomized Study of Tianjiu (Auto-moxibustion) Effects in Patients With Intradialytic Hypotension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yen Tsai, Department of TCM, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chang Gung IRB 102-4749A3
Record Dates: First submitted 2014-08-03; First posted 2014-08-06 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Intradialytic Hypotension
Keywords: Auto-moxibusition, intra-dialytic hypotension, hemodialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tianjiu (auto-moxibustion) (Experimental): The participants in the Tianjiu group will be treated with Chinese herbal patches at acupoints on the abdomen and plantar, three times per week, for 4 hours each time during HD.
  Interventions: Other: Tianjiu
- Non-Tianjiu (Non auto-MO) (Placebo Comparator): The participants in the control group will be given placebo patches (brown clay patches) on the same sites.
  Interventions: Other: Placebo (non-Tianjiu)

INTERVENTIONS:
Other: Tianjiu — After randomization, patients in Tianjiu and placebo (non-Tianjiu) groups will receive 12 sessions of treatment over a 4-week treatment period.The format of the Tianjiu intervention will be the same as in the treatment group. Participants will be instructed to lie supine before their HD session, and then the bilateral KI1 and CV4
  Other Names: auto-moxibustion, herbal acupoint paste
  Arms: Tianjiu (auto-moxibustion)
Other: Placebo (non-Tianjiu) — The format of the placebo (clay) intervention will be the same as in the treatment group.
  Arms: Non-Tianjiu (Non auto-MO)

SUMMARY:
Intradialytic hypotension (IDH) is a most frequent complication of hemodialysis (HD) and may contribute to cardiovascular events and high mortality. The etiology of IDH is multifactorial; therefore, it remains a challenging problem in the management of HD patients. Because moxibustion (MO) at specific points can influences hemodynamics, we hypothesize that Tianjiu (auto-MO) at the traditionally used meridian points will reduce the severity of hypotension in patients who undergo HD.

DETAILED DESCRIPTION:
In this clinical trial, 45 patients had IDH were divided randomly into two (auto-MO therapy and control) groups for 4 weeks. In the Tianjiu (auto-MO) group, the patients were applied at 3 points (Conception Vessel 4, and Kidney 1) for 3-4 h during HD sessions. All number of episodes complicated by symptomatic IDH during HD sessions and the number of IDH-related nursing interventions (Trendelenburg position, manual reduction of ultrafiltration rate, infusion of isotonic saline or hypertonic fluid, lowering of dialysate temperature) in a session were recorded. Pre- and post-dialysis systolic and diastolic BP, pre- and post-dialysis body weights, interdialytic weight gain, percentage of target ultrafiltration achieved, patient's subjective assessment of the degree of fatigue after dialysis (scale from 0 to 10; 0, not at all, 10, extremely) and recovery time from fatigue after dialysis were measured at the 0, 2nd, 4th and 6th week.

ELIGIBILITY:
Inclusion Criteria:

* The subjects enrolled in the study were patients undergo regular hemodialysis, ranging from 20-75 years of age, at nephrologic clinic in KCGMH. These patients have experienced > 3 episodes of intradialytic hypotension in recent two months.

Exclusion Criteria:

* (1)confounding diseases such as sepsis, cancer, decompensated liver cirrhosis, respiratory failure, and heart failure(NYHA>3), (2) disturbed consciousness, (3) pregnancy, (4) can't tolerate the heat and allergy to automoxibustion,

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The % of target ultrafiltration achieved | 1 year
  The actual ultrafiltration volume divided by the target ultrafiltration volume

SECONDARY OUTCOMES:
The frequency of IDH episodes and number of nursing interventions during HD sessions | 1 year
  The number of IDH record and related nursing intervention during each H/D session
patient's participative assessment of the degree of fatigue after dialysis (scale from 0-10) | 1 year
  The improvement of subjective symptom
Patients' recovery time from fatigue after dialysis | 1 year
  Recovery time is recorded within minutes, when arriving home, at bed time, the next morning, by next HD

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the progress to decide.

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Tsai MY, Su YJ, Ng HY, Chen SY, Huang YC, Wu CH, Chen YH. Study protocol for a single-blind, placebo-controlled randomised trial of Tianjiu effects in patients with intradialytic hypotension. BMJ Open. 2016 Mar 10;6(3):e009976. doi: 10.1136/bmjopen-2015-009976. PMID 26966058